CLINICAL TRIAL: NCT05977179
Title: A Diet Intervention Study To Mitigate Fatigue Symptoms And To Improve Muscle And Physical Function In Older Adults With Post-Acute COVID-19 Syndrome
Brief Title: Dietary Intervention to Mitigate Post-Acute COVID-19 Syndrome
Acronym: Long-COVIDiet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Galya Bigman, Assistant Professor, University of Maryland, School of Medicine, Baltimore, MD, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HP-00106745
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Post-Acute COVID-19 Syndrome; Fatigue
Keywords: COVID; long-COVID; DIET
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary intervention to mitigate Post-Acute COVID-19 Syndrome (Experimental): During the intervention, participants will receive an individual dietary plan from a Registered Dietitian (RD) that emphasizes nutrients with high anti-inflammatory activity, which can be obtained from various foods and supplements (e.g., vitamin D, omega-3, and quality protein). Additionally, participants will actively participate in weekly dietary sessions that cover topics from 'What's On Your Plate?', specifically tailored to address the nutrition recommendations for older adults in the Dietary Guidelines for Americans 2020-2025.
  Interventions: Other: Dietary intervention to mitigate Post-Acute COVID-19 Syndrome
- Attention Control (Other): Participants in the control group will receive an equal amount of social attention, in terms of both dose and duration, comparable to that provided in the intervention group. Topics covered during these sessions will focus on healthy aging, including oral health, hearing loss, eyesight, and ensuring a safe environment by addressing issues such as gas leaks, fire hazards, and fall prevention. No dietary information will be included in these discussions.
  Interventions: Other: Attention Control

INTERVENTIONS:
Other: Dietary intervention to mitigate Post-Acute COVID-19 Syndrome — As it was described in the arm/group descriptions.
  Arms: Dietary intervention to mitigate Post-Acute COVID-19 Syndrome
Other: Attention Control — As it was described in the arm/group descriptions.
  Arms: Attention Control

SUMMARY:
The primary objective of this study is to conduct a 16-week randomized controlled trial aimed at investigating the effectiveness of the Whole-Diet Approach when following a healthy US-style diet rich in anti-inflammatory properties. The study will focus on evaluating its impact on reducing symptoms related to Post-Acute Sequelae of SARS-CoV-2 Infection (PACS) in adults aged 50 years and older.

The main research questions this study aims to answer are:

1. Does adhering to a healthy US-style diet, which is abundant in anti-inflammatory properties, effectively mitigate fatigue symptoms in adults with PACS?
2. Does adhering to a healthy US-style diet, which is abundant in anti-inflammatory properties, effectively mitigate declines in muscle function and physical performance in adults with PACS?

At the beginning of the study, eligible participants will be randomly assigned to either the Dietary Intervention Group, where they will receive personalized dietary plans and weekly sessions, or the Attention Control Group, where they will attend general health sessions on a weekly basis as well.

This research intends to shed light on the potential benefits of the Whole-Diet Approach and its role in ameliorating PACS-related symptoms among older adults. By comparing the outcomes of the two groups, we hope to gain valuable insights into the effectiveness of this dietary intervention in improving the quality of life for individuals dealing with PACS.

DETAILED DESCRIPTION:
The main objective of this research is to evaluate the impact of the 'Whole-Diet Approach' through a 16-week randomized-controlled dietary intervention on reducing symptoms of PACS (Post-Acute Sequelae of SARS-CoV-2 Infection), specifically targeting fatigue and muscle weakness.

The study will include 56 men and women aged 50 years or older, all diagnosed with PACS. These participants will be randomly assigned to one of the two groups:

1. Dietary Intervention Group: Participants in this group will benefit from a personalized dietary plan created by a skilled Registered Dietitian (RD). The dietary recommendations will align with the U.S. Healthy diet style as outlined by the Dietary Guidelines for Americans 2020-2025. Weekly group sessions with the RD/Principal Investigator (PI) will facilitate the practical application of the personalized diet. The RD will also focus on promoting the intake of foods with high anti-inflammatory activities.
2. Attention Control Group: Participants in this group will attend educational sessions on general health topics, such as healthy aging (e.g., oral health, hearing loss, eyesight) and safety environment (e.g., gas leaks, fire, fall hazards). However, they will not receive any specific dietary information.

Throughout the 16-week intervention period, all participants will be required to strictly adhere to their prescribed dietary plan and attend the designated sessions.

The study's primary objectives are as follows:

Aim 1: Evaluate the effect of the Whole-Diet Approach on the participants' Healthy Eating Index and fatigue levels, in comparison to the attention control group, among adults with PACS.

Aim 2: Assess the impact of the dietary intervention on muscle mass, strength, and physical function in adults with PACS, and compare these outcomes with the attention control group.

By addressing these key aims, this research will provide valuable insights into the effectiveness of the Whole-Diet Approach as a potential intervention for alleviating symptoms related to PACS and enhancing overall well-being among older adults.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 50 years or older
2. No known active infectious disease (COVID-19 or other).
3. Participant diagnosed with long-COVID/ post- acute COVID-19 syndrome (PACS) /ICD-10-CM codes U09.9
4. Moderate/severe fatigue Brief Fatigue Inventory (BFI)≥4
5. Poor diet quality assessed by the short Healthy Eating Index (HEI)<70

Exclusion Criteria:

1. Participants with a home oxygen requirement or requiring chronic ventilator support
2. Participants diagnosed with diabetes who do not have a recent HbA1c level or with HbA1c > 9%
3. Participants diagnosed with Congestive Heart Failure (CHF New York Heart Association) > class 2
4. Participants with dietary restrictions due to medication use that affects blood clotting, such as Warfarin or other reasons.
5. Evidence of any condition as determined by a physician or the study team that would lead to an increased risk of illness due to any aspect of proposed testing and interventions, or introduce unanticipated confounding of study results.
6. Participants diagnosed with uncontrolled hypertension that will be defined as:

   1. Systolic blood pressure consistently equal to or higher than 190 mmHg.
   2. Diastolic blood pressure consistently equal to or higher than 110 mmHg.
   3. Participants with a recent history of hypertensive crisis (severe elevation in blood pressure requiring immediate medical intervention), regardless of current blood pressure levels.
7. Participants with diet restrictions or allergies that can affect adherence to the diet, such as allergy to fish or shellfish.
8. Participation in another trial in which active intervention is being received.
9. Participants with active drug or alcohol use/dependence that would interfere with adherence to the study.
10. Participants scheduled for surgical procedures within the next 6 months.
11. Participants diagnosed with active cancer.
12. Participants diagnosed with liver diseases.
13. Participants diagnosed with kidney-related conditions, including Chronic Kidney Disease (CKD) > stage 3.
14. Below the age of 50 years.

Ages: 50 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue | Baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks (end of the trial)
  Fatigue will be assessed by the brief fatigue inventory (BFI)
Physical Function | Baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks (end of the trial)
  Physical Function will be measured by the Short Physical Performance Battery(SPPB)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No